CLINICAL TRIAL: NCT06950554
Title: From Clinic to Smartphone: Evaluating the i-TUG for Balance and Fall Risk in Chronic Stroke
Brief Title: Validity and Reliablity of i-TUG Via EncephaLog
Acronym: EncephaLog
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Merve SEVINC GUNDUZ, RESEARCH ASSISTANT, Bezmialem Vakif University
Other Study IDs: 12.11.2024-171654
Record Dates: First submitted 2025-04-18; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Stroke, Ischemic; Balance Assessment; Smartphones
Keywords: Stroke, Balance, Berg balance scale, Rehabilitation, EncephaLog
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EncephaLog Assessment Group: The EncephaLog is an FDA-cleared, smartphone-based application designed to assess dynamic balance and gait disorders in older adults and individuals with neurological or non-neurological conditions. The application uses the smartphone' built-in accelerometer and gyroscope to deliver reliable and valid kinematic assessments.

SUMMARY:
This study investigated the test-retest reliability and construct validity of the i-TUG, standard TUG, and Berg Balance Scale (BBS) using the EncephaLog smartphone application in individuals with chronic ischemic stroke. A total of 49 participants were assessed in two sessions to evaluate test-retest reliability. Construct validity was analyzed using Pearson correlation coefficients. Standard Error of Measurement (SEM) and Minimal Detectable Change (MDC) values were also calculated.

DETAILED DESCRIPTION:
The study was conducted with 37 individuals diagnosed with chronic ischemic stroke. Participants were assessed using the i-TUG, TUG, BBS, and additional postural sway parameters collected via EncephaLog. Two test sessions were conducted to assess test-retest reliability. Pearson correlation coefficients were used to evaluate construct validity, and the Standard Error of Measurement (SEM) and Minimal Detectable Change (MDC) were also calculated.

Inclusion Criteria:

* voluntary participation,
* a diagnosis of stroke, no involvement in any physiotherapy program for at least three months prior to the study,
* age between 18 and 75 years,
* the ability to walk independently Functional Ambulation Scale (FAS) score greater than 3,
* the spasticity of the m. gastrocnemius was graded as 2 or less on the Modified Ashworth Scale (MAS).

Exclusion Criteria:

* severe visual or cognitive impairments,
* severe cardiovascular disease, or musculoskeletal conditions or skin disorders that affected the lower extremities.

ELIGIBILITY:
Inclusion Criteria:

voluntary participation, a diagnosis of stroke, no involvement in any physiotherapy program for at least three months prior to the study, age between 18 and 75 years, the ability to walk independently Functional Ambulation Scale (FAS) score greater than 3, and the spasticity of the m. gastrocnemius was graded as 2 or less on the Modified Ashworth Scale (MAS).

Exclusion Criteria:

Participants were excluded if they had severe visual or cognitive impairments, severe cardiovascular disease, or musculoskeletal conditions or skin disorders that affected the lower extremities.

Ages: 18 Days to 75 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ischemic stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
Instrumental Timed Up and Go Test (i-TUG) by EncephaLog | Day 1 and Day 7
  The EncephaLog is an FDA-cleared, smartphone-based application designed to assess dynamic balance and gait disorders in older adults and individuals with neurological or non-neurological conditions. The application uses the smartphone' built-in accelerometer and gyroscope to deliver reliable and valid kinematic assessments.
Timed Up and Go Test (TUG) | Day 1 and Day 7
  The TUG test is a commonly used and validated measure to assess balance and mobility. Initially developed for older adults, 29 it has since been widely adopted for neurological and pediatric populations. 30-32 The test requires the participant to rise from a chair, walk 3 meters, turn, return, and sit down. The time to complete the task is recorded. A score greater than 13.5 seconds indicates an increased risk of falling in elderly.
Berg Balance Scale (BBS) | Day 1 and Day 7
  The BBS consists of 14 items designed to assess postural control and fall risk in elderly individuals. 35 Tasks include sitting to standing, standing unsupported, transfers, turning, and stepping. Each item is scored from 0 to 4, and the total score ranges from 0 to 56. A score between 0-20 indicates high fall risk and need for assistive devices; 21-40 indicates moderate fall risk; and 41-56 indicates low fall risk with no need for assistive devices.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Eyupsultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified data (i-TUG, TUG, and BBS scores) will be available upon request after publication for research purposes.
Supporting Information: Study Protocol, Analytic Code
Time Frame: De-identified individual participant data and supporting documents (study protocol, statistical analysis plan, and analytic code) will be available beginning 6 months after publication and will remain available for 2 years.
Access Criteria: Qualified researchers affiliated with academic institutions will be able to request access to de-identified individual participant data (i-TUG, TUG, BBS scores), study protocol, statistical analysis plan, and analytic code. Requests should be submitted to the corresponding author and will be reviewed by the study team. Data will be shared via secure institutional data transfer platforms.